CLINICAL TRIAL: NCT06877832
Title: Determinants of Acute Effects of Stretching Vs. Foam Rolling: Morphological, Sensory and Fluid Responses
Brief Title: Effects of Foam Rolling, Foam Rolling with Dynamic Movement, and Static Stretching on Plantar Flexor Range of Motion and Tissue Properties in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewan Thomas (Other)
Responsible Party: Sponsor-Investigator, Ewan Thomas, Professor, University of Palermo
Organization: University of Palermo (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 170/2023
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Healthy Subjects (HS)
Keywords: stiffness; jump; pain sensitivity; EIM; L-BIA
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Static Stretching (SS) (Experimental): For the SS, participants will be instructed to stand and place their dominant foot on a wedge with a 35° incline. They will stretch the plantar flexor muscles for 30 seconds, performing 4 repetitions.
  Interventions: Other: Static Stretching (SS)
- Foam Rolling (FR) (Experimental): For the FR, participants will be instructed to position the muscle belly of the PF on the roller. Thirty rolls (15 proximal and 15 distal) for a duration of 30 seconds will be considered one set.
  Interventions: Other: Foam Rolling (FR)
- Foam Rolling with Dynamic Movement (FR-DM) (Experimental): The FR-DM will involve positioning the muscle belly of the PF on the roller and, without moving the roller, performing 15 plantar flexions and 15 dorsiflexions of the ankle for a period of 30 seconds while compressing the dominant leg with the contralateral leg.
  Interventions: Other: Foam rolling with dynamic movement (FR-DM)
- Control Group (CG) (No Intervention): The CG will only perform the assessment tests, remaining seated for 4 minutes between the pre-test and post-test.

INTERVENTIONS:
Other: Static Stretching (SS) — For the SS, participants will be instructed to stand and place their dominant foot on a wedge with a 35° incline, stretching the plantar flexor muscles.
  Arms: Static Stretching (SS)
Other: Foam Rolling (FR) — For the FR, participants will be instructed to position the muscle belly of the PF on the roller. Thirty rolls (15 proximal and 15 distal) will be performed on the muscle belly while maintaining compression on the muscle.
  Arms: Foam Rolling (FR)
Other: Foam rolling with dynamic movement (FR-DM) — The FR-DM will involve positioning the muscle belly of the PF on the roller and, without moving the roller, performing 15 plantar flexions and 15 dorsiflexions of the ankle for a period of 30 seconds while compressing the dominant leg with the contralateral leg.
  Arms: Foam Rolling with Dynamic Movement (FR-DM)

SUMMARY:
Each voluntary participant will be invited and tested at the Functional Assessment Laboratory. After reading and completing the informed consent document regarding our research and data processing, participants will be invited for four separate sessions at the laboratory. During the first session, essential personal information (name, surname, sex, age) will be recorded. Immediately after measuring the participant's height using a stadiometer and weight using a scale, several tests will be conducted to assess pain thresholds and tissue density using specific dynamometers, joint mobility levels of the participants (Passive Muscle Mobility Test and a test using the accelerometer), and a Bioimpedance Analysis to assess body fluids. After a 15-minute rest period, the tests will be repeated to obtain an initial baseline control assessment. The subsequent sessions will involve the same evaluations, which will be conducted before, immediately after, and 15 minutes after the proposed intervention. The proposed interventions will be randomized across the sessions and will alternatively include: a brief session of static stretching on the leg muscles (4 sets of 30 seconds with 15 seconds of rest between sets), a session of static foam rolling (4 sets of 30 seconds with 15 seconds of rest between sets) on the same muscle groups, where pressure is applied to the muscle through the participant's body weight on a foam roller while performing muscle contractions, or dynamic foam rolling, during which the muscle will be rolled over the foam roller.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants, adult participants, active, agreeing to sign the consent form

Exclusion Criteria:

Participants with neuromuscular, orthopedic and gynecological disease (or taking oral contraceptives) or those having injuries of the lower extremities were excluded from the investigation. Female participants were allowed to participate to the experiments only during the follicular phase of their menstrual cycle and always before ovulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Plantar Flexors ROM | 5 minutes
  Each participant was placed prone on a medical bed with both feet hanging out of the bed. Inelastic straps were used to fix the pelvis and the contralateral leg of the tested participant. A flat rigid surface was fixed on the sole of the foot. A two arm electronic goniometer (Digital Angle Ruler, resolution0.05°, accuracy±0.2°, repeatability0.05°) was then placed with one arm parallel to the flat surface positioned on the foot sole and the other arm following the diaphysis of the fibula. Starting position was set with the foot and the leg forming a 90°angle. The investigator passively pushed the foot into a dorsiflexion motion to the limit of available ROM, or the maximum tolerable pain for each participant.
Pain Pressure Thresholds | 5 minutes
  PPT was assessed through a portable algometer(FPX25 Pain Tester, Wagner Instruments,CT,USA). The participant's measurement position and posture were similar to TH. The algometer was positioned perpendicular to the direction of the muscle fibers. The investigator pushed the metal rod of the algometer at a pressure of 1kg per second over the muscle belly of the participant. The participant was instructed to say "stop" when pain, rather than just pressure, was experienced.
Localised Bioimpedance Analysis (L-BIA) | 5 minutes
  L-BIA was performed using a single frequency phase-sensitive device(BIA-101 Anniversary Sport Edition, Akern Systems, Firenze-Italy) at 50kHz and 400μA to measure PhA and vector length. Two pairs of electrodes (source(I) and detector(V) electrodes) were used. One pair was positioned on the upper part of the leg, with the lateral part of the I positioned on the popliteal crease(Lee et al., 2023) and the V, positioned caudally, parallel to I, 5cm apart. The other pair was positioned on the lower part of the leg with the lateral part of the I positioned above the tibial malleolus and the V, in a cranial direction parallel to I, 5cm apart. Prior to each test, the BIA measurements of the analyzer were validated using a precision circuit with acceptance for resistance(R) measurements of 383ohm(Ω) and reactance(Xc) values of 45Ω.
Drop Jump Height (DJ) | 5 minutes
  A unilateral DJ was assessed through an Optojump™ system(Microgate, Bolzano, Italy) connected to a personal computer with dedicated software(OptojumpTM Next software). The system consists of two optical bars, a receiver and a transmitter, positioned 1m apart. The bars identify ground contact time(with a precision of 1ms) and then convert non-contact time into cm. Based on recommendations on optimal jump height(20 to 60cm), all jumps were performed from a box with a height of 40cm. Participants had to stand upright on the box with their hands positioned on their hips. At the "go" of the investigator, the participants had to jump forward from the box into the opto-jump system avoiding stepping down from the box or hopping off of the box. Once the participant reached the ground with their dominant limb, without flexing the knee, had to jump as high as possible. A 30s rest was given between each trial.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Palermo, Palermo, PA, Italy

IPD SHARING:
Plan to Share IPD: No